CLINICAL TRIAL: NCT01496547
Title: Sequential Intensive Chemotherapy Followed by Allogeneic Stem Cell Transplantation With Reduce-intensity Conditioning for Refractory and Relapse Acute Myeloid Leukemia in Adult Patients
Brief Title: Sequential Intensive Chemotherapy Followed by RIC for Refractory and Relapse AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-2011-RefactoryAML-SCT
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2016-05

CONDITIONS: Acute Leukemia
Keywords: feasibility, effective and safety; intensive chemotherapy; RIC regimen; refractory or relapse leukemia; allogeneic stem cell transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intensive chemo - RIC preparation (Experimental): The intensive chemotherapy is composed of Fludarabine 35mg/m2 D1-5, high-dose cytarabine 2g/m2 D1-5 + idarubicin (12mg/m2) D5-7. The reduced intensity preparation regimen will start 7 days after the chemotherapy with fludarabine 35mg/m2 for 5 days + iv busulfan 3.2mg/kg/day for 3 days followed by stem cell infusion 2 days later.
  Interventions: Drug: intensive chemo - RIC preparation

INTERVENTIONS:
Drug: intensive chemo - RIC preparation — The intensive chemotherapy is composed of fludarabine 35mg/m2 + high-dose cytarabine 2g/m2 D1-5 + idarubicin (12mg/m2) D5-7. The reduced intensity preparation regimen will start 7 days after the chemotherapy with fludarabine 35mg/m2 for 5 days + iv busulfan 3.2mg/kg/day for 3 days followed by stem cell infusion 2 days later.
  Other Names: FLAG-IDA-RIC

SUMMARY:
Patients with refractory and relapse leukemia had poor outcome even with allogeneic stem cell transplantation. In our previous retrospective study, the overall survival is 14.6+/-8.8% while 90% patients eventually relapsed with marrow ablative conditioning mostly standard iv-Bu-Cy or Cy-TBI. The accumulated TRM is 29.5+/-11.5%. Thus our data suggested that the conventional transplantation approach may not be able to overcome the refractory disease. A new strategy to combined a low dose regimen following intensive chemotherapy for tumor reduction seems to be effect in both relapsed. high-risk and refractory AML or ALL. In this study, we focus on a new treatment strategy for particular refractory AML patients.

DETAILED DESCRIPTION:
This is a single arm phase II trial to test the efficacy and feasibility of new sequential intensive chemo and transplantation approach for refractory leukemia. Patients with refractory acute myeloid or lymphoblastic leukemia are enrolled in this trial. Patients will received intensive chemotherapy including Fludarabine, cytarabine and idarubicin as (FLAG-IDA). Seven days after the chemotherapy, sequential transplantation conditioning regimen as fludarabine and busulfan will be given.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with refractory or relapse acute myeloid leukemia not in remission after 2 cycles of induction chemotherapy early relapse (1st remission less than 6 months) not in remission after 1 cycle of re-induction chemotherapy multiple relapse
* age 16-60 years
* with inform consent
* no contraindication for allogeneic transplantation: active infection, allergy to FLu/Bu/CTX, liver and renal function damage
* HLA matched related (6/6) or unrelated donors (at least 8/10)

Exclusion Criteria:

* age less than 18 years or over 61 years
* liver function/renal function damage (over 2 X upper normal range)
* with mental disease

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2018-02-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2-year

SECONDARY OUTCOMES:
non-relapse mortality | 2-year
relapse rate | 2-year
overall survival | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang W, Fan X, Wang L, Hu J. Busulfan and fludarabine conditioning regimen given at hematological nadir of cytoreduction fludarabine, cytarabine, and idarubicin chemotherapy in patients with refractory acute myeloid leukemia undergoing allogeneic stem cell transplantation: a single arm pilot consort study. Medicine (Baltimore). 2015 Apr;94(15):e706. doi: 10.1097/MD.0000000000000706. PMID 25881847